CLINICAL TRIAL: NCT03094585
Title: Nurses Knowledge About and Attitude Towards Clinical Trials. A Randomised Trial
Brief Title: The INFO-II Trial: Nurses Knowledge About and Attitude Towards Clinical Trials
Acronym: INFO-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Collaborators: Section for Health Services Research, Department of Public Health, Copenhagen University Hospital (Unknown); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Protocol: 1996-10-31/KK.df; 1997-DP-31-RKF-5-INFO-II [CTU]
Record Dates: First submitted 2016-08-25; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Healthy nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No information (No Intervention): The nurses in this group are offered no booklet or oral information
- Written and oral information (Experimental): The nurses in this group are offered written information which consisted of a booklet describing basic aspects of clinical research including aim, background, formalities, ethics, informed consent, randomisation, blinding, placebo, drug development, and financial aspects. Furthermore, they are offered oral information which consisted of group sessions focusing on active feedback
  Interventions: Other: Written and oral information
- Written information (Experimental): The nurses in this group are offered written information which consisted of a booklet describing basic aspects of clinical research including aim, background, formalities, ethics, informed consent, randomisation, blinding, placebo, drug development, and financial aspects.
  Interventions: Other: Written information

INTERVENTIONS:
Other: Written and oral information — The written information (booklet) was 12 A4 pages long and took about 15 minutes to read. The oral information consisted of group sessions which focused on active feedback. Each session was lead by one of the authors who first went through the topics described in the booklet. The review of the topics was followed by a plenary discussion.
  Arms: Written and oral information
Other: Written information — The written information (booklet) was 12 A4 pages long and took about 15 minutes to read.
  Arms: Written information

SUMMARY:
The purpose of this study is to examine (a) nurses' knowledge about and attitude towards clinical research, and (b) the effect of written and oral information on nurses' knowledge about and attitude towards clinical research.

DETAILED DESCRIPTION:
A randomised (1:1:1), evaluator-blinded educational trial on written and oral information versus oral information alone versus no information on nurses' knowledge about and attitude towards clinical research in a university hospital in Copenhagen, Denmark. The investigators planned to randomise 213 nurses (approximately 71 to each intervention group) based on a minimal relevant difference of 1.6 points on the knowledge scale, a standard deviation of 3.1 points, a beta (type II error) risk of 0.20, and an alpha of 0.025. At entry and two weeks later, the nurses should complete two validated questionnaires, which indicated their knowledge on a 0-17 point scale and their attitude on a 0-156 point scale. Predictors of the entry knowledge and attitude and changes in knowledge and attitude after interventions were planned to be identified through adjusted ANOVA. The effects of the active interventions were compared with the control and adjusted for multiple comparisons. Interventions: Written and oral information: The nurses in this group are offered the written information consisted of a booklet which described basic aspects of clinical research including aim, background, formalities, ethics, informed consent, randomisation, blinding, placebo, drug development, and financial aspects. The booklet was developed with the assistance of nurses, physicians, psychologists, researchers, and communication experts. The booklet was adjusted after repeated pilot tests among laymen and employees at our research institution. The booklet was 12 A4 pages long and took about 15 minutes to read. In the INFO I trial, the booklet had a significant effect on outpatients' knowledge about and attitude towards clinical research. The oral information consisted of group sessions which focused on active feedback. Each session was lead by one of the authors who first went through the topics described in the booklet. The review of the topics was followed by a plenary discussion. The sessions lasted 15 to 40 minutes, depending on the interest of the nurses. Written information: The nurses in this group are offered the written information consisted of the same booklet as above, but without oral information. No information: The nurses in this group are offered no booklet or oral information.

ELIGIBILITY:
Inclusion Criteria:

* Graduated nurse
* Signed informed consent

Exclusion Criteria:

* Participant in another trial similar to the present trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1997-09; Primary Completion 1997-09 (Actual)

PRIMARY OUTCOMES:
Knowledge score (questionnaire) | Two weeks
  The primary outcome is obtaining satisfactory knowledge score by using a Knowledge questionnaire.

SECONDARY OUTCOMES:
Attitude towards clinical research and randomized clinical trials (questionnaire) | Two weeks
  Secondary outcome is the attitude towards clinical research and randomized clinical trials. This is obtained by using a attitude questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Krogsgaard, MD, Principal Investigator — Copenhagen Trial Unit - Centre for Intervention Research, Denmark
Locations (2):
- Denmark (2):
  - Copenhagen Trial Unit, Centre for clinical intervention research, Coepnhagen
  - Hvidovre University Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No
No plan for data sharing